CLINICAL TRIAL: NCT05591859
Title: Restoration Anatomic Acetabular Shell Revision Study - A Post-market, Multi-center Evaluation of the Clinical Outcomes of the Restoration Anatomic Acetabular Shell in a Revision Indication
Brief Title: Restoration Anatomic Acetabular Shell Revision Study
Acronym: RAS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stryker Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 105
Record Dates: First submitted 2022-10-19; First posted 2022-10-24 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Arthropathy; Hip Arthropathy; Hip Osteoarthritis
MeSH Terms: conditions — Joint Diseases; Osteoarthritis, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Restoration Anatomic Acetabular Shell (Other)
  Interventions: Device: Restoration Anatomic Acetabular Shell

INTERVENTIONS:
Device: Restoration Anatomic Acetabular Shell — Multi-hole acetabular shell intended for cementless fixation into a prepared acetabulum and is a modular component design that is assembled intra-operatively.

SUMMARY:
This study will be a non-randomized, ambidirectional (retrospective and prospective) study where all subjects will be followed prospectively. The study will evaluate the survivorship of the RAS acetabular component in a previously failed total hip arthroplasty (THA) in a consecutive series of subjects who meet the eligibility criteria.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a candidate for a revision of a failed acetabular component with the Restoration Anatomic Acetabular Shell.
* Subject has signed an IRB-approved, study specific Informed Consent Form (ICF).
* Subject is skeletally mature.
* Subject is a male or non-pregnant female.
* Subject is willing and able to comply with postoperative scheduled clinical evaluations.

Exclusion Criteria:

* Subject has a non-Stryker retained stem at the time of study device implantation.
* Subject has a Body Mass Index (BMI) > 45.
* Subject has an active or suspected latent infection in or about the affected hip joint at time of study device implantation.
* Subject has a mental or neuromuscular disorder which would create an unacceptable risk of prosthesis instability, prosthesis fixation failure, or complications in postoperative care.
* Subject has compromised bone stock which cannot provide adequate support and/or fixation to the prosthesis.
* Subject is diagnosed with a systemic disease (e.g. Lupus Erythematosus) or a metabolic disorder (e.g. Paget's Disease) leading to progressive bone deterioration.
* Subject is immunologically suppressed or receiving steroids in an excess of normal physiological requirements (e.g. > 30 days).
* Subject has a known sensitivity to device materials.
* Subject is a prisoner.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2024-03-02 (Actual); Primary Completion 2036-03-01 (Estimated); Study Completion 2036-03-01 (Estimated)

PRIMARY OUTCOMES:
Success rate | 10 years
  Success rate is defined as no incidence of revision for aseptic loosening

SECONDARY OUTCOMES:
Adverse Events | 10 years
  All protocol defined adverse events as well as all-cause revision and/or removal of RAS

CONTACTS AND LOCATIONS:
Locations (1):
- Regents of the University of Colorado, Denver, Colorado, United States